CLINICAL TRIAL: NCT05722652
Title: CONFIDENCE: A Pilot Randomized Control Trial With Waitlist Condition to Test a Multicomponent Clinic-based Intervention to Promote COVID-19 Vaccine Intention and Uptake Among Diverse Youth and Adolescents
Brief Title: A Multicomponent Clinic-based Intervention to Promote COVID-19 Vaccine Intention and Uptake Among Diverse Youth and Adolescents
Acronym: CONFIDENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Baystate Health (Other)
Responsible Party: Principal Investigator, Stephenie Lemon, Professor and Chief of the Division of Preventive and Behavioral Medicine, Department of Population and Quantitative Health Sciences, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00000728
Record Dates: First submitted 2023-02-08; First posted 2023-02-10 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: COVID-19 Vaccination
Keywords: Vaccination hesitancy
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Confidence Intervals

STUDY DESIGN:
Intervention Model Description: The investigators will be using a cluster, randomized control trial design, in which clinics are assigned to either the intervention or control group. Clinics in the control group or "waitlist" condition, will receive the intervention approximately 12 months later.
Who Masked: Participant
Masking Description: Clinics will know if they are assigned to the intervention or control condition. However, individual participants (parents of children ages 5 to 17) will not know if their clinic is in the intervention or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental)
  Interventions: Behavioral: CONFIDENCE
- Waitlist Condition (Active Comparator): Clinics in this condition will receive the intervention approximately 12 months after the intervention condition.
  Interventions: Behavioral: CONFIDENCE

INTERVENTIONS:
Behavioral: CONFIDENCE — This clinic-based, multicomponent intervention consists of 3 parts:
  1. Webinar training for clinicians and clinic staff about how to communicate with vaccine-hesitant parents
  2. Parent-facing educational materials about COVID-19 vaccination
  3. Support in creating a personalized poster campaign featuring providers and clinic staff sharing personal stories about COVID-19 vaccination

SUMMARY:
The goal of this study is to refine and test CONFIDENCE, a multi-component clinic-based intervention in pediatric or family practice clinical settings. Using a randomized control trial design, the investigators will assess preliminary effectiveness of the intervention to increase COVID-19 vaccine intention among parents of under-vaccinated children ages 5 to 17.

Participating clinics will receive a brief intervention consisting of: (1) webinar training focused on communication with vaccine-hesitant parents, (2) parent-facing educational materials about COVID-19 vaccination, (3) support to create a personalized, poster campaign featuring providers. Clinics in the control condition will receive the intervention approximately 12 months after the clinics in the intervention condition.

ELIGIBILITY:
Practice site inclusion criteria

* Pediatric or family practice clinic that serves pediatric population (ages 5 to 17)
* Affiliated with UMass Memorial Health Care and/or Baystate Health
* Serve a patient population that is at least 30% racial/ethnic minority group members.

Inclusion Criteria for Parents:

The following inclusion criteria will be applied to parents (on behalf of their children):

* Parent/guardian (referred to as parents in this proposal) of child between ages 5 and 17
* Able to read and write in English, Spanish, Portuguese or Vietnamese, which are the predominant languages in the target communities
* Parent of patient at participating clinical site/child received non-urgent care visit during study period
* Child not up-to-date for COVID-19 per current CDC guidelines at the time of enrollment.

Exclusion Criteria for Parents:

°Parent under age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
COVID-19 vaccine intention | Data collection will occur in the four weeks following implementation
  Parent exit survey in clinics: Parents will report their intention to vaccinate their children for COVID-19. See survey question below:
  "Did you decide to vaccinate your child against COVID-19 today? Yes/No"

SECONDARY OUTCOMES:
Feasibility: Recruitment | End of study; approximately 15 months
  Completion of the parent exit surveys will be documented and used to calculate the percentage of eligible parents (those who received a form) who completed the survey.
Feasibility: Data Completeness | End of study; approximately 15 months
  Data completeness/missing data for all participant-level measures from the parent exit survey at the item-level will be examined. An exploratory analysis will be conducted to further decipher the quality of COVID-19 vaccination data in electronic medical records to determine its potential utility in a future trial.
Feasibility: Randomization | End of study; approximately 15 months
  Recruitment, data completion and participant characteristics will be compared across the two study conditions to determine if differences emerge.
Acceptability: Parents | Four to eight weeks post implementation
  Perceived acceptability will be assessed via the survey question "How satisfied were you with the conversations about COVID-19 vaccination for your child at your visit today", which will have a 3-point Likert response scale, ranging from not at all to very satisfied.
Perceived appropriateness: Parents | Four to eight weeks post implementation
  Perceived appropriateness will be assessed via the survey question "How appropriate were the conversations about COVID-19 vaccination for your child at your visit today?"
Implementation Fidelity | Four to eight weeks post implementation
  Implementation fidelity will be assessed by three questions that ask about provider's behavior regarding the intervention: "Did you and the provider discuss COVID-19 vaccination for your child today?"; "Did the provider share their own COVID-19 experience with you?"; and "Did the doctor give you any materials about the COVID-19 vaccination today?".
Acceptability: Providers and clinic staff | Four to eight weeks post implementation
  Will be assessed qualitatively through semi-structured interviews using questions like "How satisfied were you with intervention activities?"
Perceived Appropriateness: Providers and clinic staff | Four to eight weeks post implementation
  Will be assessed qualitatively through semi-structured interviews using questions like "How relevant were intervention components and how compatible was the intervention with values and the workflow of the practice?"
Perceived feasibility: Providers and clinic staff | Four to eight weeks post implementation
  Will be assessed qualitative through semi-structured interviews using questions like "What is the likelihood of sustaining the implementation of the intervention component in practice after the research study concludes."

CONTACTS AND LOCATIONS:
Overall Officials: Stephenie C Lemon, PhD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified individual-level dataset will be made available to researchers who make a reasonable request to the principal investigator. Data will be made available upon publication of the primary outcomes manuscript.
Time Frame: Data will be available will be available upon publication of the primary outcomes manuscript from this project.
Access Criteria: Data will be made available upon reasonable request from researchers.

REFERENCES:
- [Background] Ryan GW, Goulding M, Borg A, Minkah P, Beeler A, Rosal MC, Lemon SC. Development and Beta-Testing of the CONFIDENCE Intervention to Increase Pediatric COVID-19 Vaccination. J Pediatr Health Care. 2023 May-Jun;37(3):244-252. doi: 10.1016/j.pedhc.2022.11.002. Epub 2022 Nov 17. PMID 36470798